CLINICAL TRIAL: NCT04952025
Title: Brain Imaging Study of Amyotrophic Lateral Sclerosis Based on Accurate Brain Volume Quantitative Analysis
Brief Title: Quantitative Analysis of Precise Brain Volume in Amyotrophic Lateral Sclerosis
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: M2020369
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALS patients
  Interventions: Diagnostic Test: Diagnostic criteria
- normal controls

INTERVENTIONS:
Diagnostic Test: Diagnostic criteria — Diagnostic criteria of ALS
  Groups: ALS patients

SUMMARY:
Using the original MRI images of 16 ALS patients and 16 normal controls matched by gender, age and education level in the previous study, the differences of brain volume in different parts of ALS patients and normal controls, and the correlation between brain structure and clinical characteristics were compared by precise brain volume quantitative analysis technology.

DETAILED DESCRIPTION:
This study was a retrospective study. The subjects were 16 ALS patients and 16 normal controls. Previous studies have collected patients' age, gender and education level; The onset site, onset time, bulbar involvement, diagnostic grade, ALSFRS-R score, application of ventilator, application of lirutai, gastrostomy; Age, gender and education level were collected in the control group. Accurate quantitative analysis of brain volume was performed on the original brain MRI images of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed ALS patients
* healthy volunteers

Exclusion Criteria:

* none

Age Groups: Child, Adult, Older Adult
Study Population: 32
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Accurate quantitative analysis of brain volume | 1 day
  Accurate quantitative analysis of brain volume using magnetic resonance brain imaging

SECONDARY OUTCOMES:
general situation | 1 day
  Age, gender and education level were collected; Onset site, onset time, involvement of bulbar, diagnostic grade, ALSFRS-R score, application of ventilator, application of lirutai, gastrostomy

CONTACTS AND LOCATIONS:
Overall Officials: Shan Ye, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No